CLINICAL TRIAL: NCT06420167
Title: DapagliFLOzin in Renal AL Amyloidosis (FLORAL)
Acronym: FLORAL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Jeffrey Zonder, Principal Investigator, Multiple Myeloma Multidisciplinary team leader, M.D., Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-074
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Renal AL Amyloidosis
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dapagliflozin (Experimental): Dapagliflozin 10mg orally, daily for 6 months
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — 10mg orally once daily
  Other Names: BMS-512148; Forxiga® / Farxiga®

SUMMARY:
The goal of this clinical trial is to learn if an oral drug called dapagliflozin is safe and can reduce high protein levels in the urine of patients with renal amyloid light-chain (AL) amyloidosis using a decentralized study design.

Participants will be:

* screened for the trial via an online platform
* contacted by study personal to obtain electronic consent
* enrolled in the trial if eligible and consented
* contacted by study personal for further instructions and directions
* sent dapagliflozin oral medication (supplied by the site pharmacy)
* followed up regularly with the study team via telemedicine or other online avenues
* monitored using lab work, inquiries about side effects and assessment of protocol adherence at 1 month, 3 months and 6 months
* continue treatment for 6 months

DETAILED DESCRIPTION:
1. Participants are recruited by one of the following methods:

   1. Self-referral through the website
   2. Receiving recruitment materials from their provider.
2. Participant visits the prescreening website.

   1. High level prescreening questions are answered by the participant.
   2. If appropriate based on answers to the questions, the participant may provide their contact information for follow up by the study team.
3. Study team contacts potential participants to review the study and explain next steps
4. Participant is provided with the link and password to view the video and sign the consent via Adobe Sign
5. An investigator will meet virtually with the participant to obtain medical history information, concomitant medications, and performance status (screening visit)
6. Once the participant passes screening in step 5, an order will be sent to the participant for the remaining screening labs to be done at a local laboratory that is covered by their insurance
7. The lab will fax results to the site
8. After review of eligibility and the study team will proceed with enrolling the participant if appropriate
9. The participant will proceed to the baseline visit (telehealth for any portion that can be done via phone/video and order for lab tests as previously described) if needed to comply with the protocol calendar/window.
10. The participant is approved to begin dosing by the investigator
11. The site will dispense via mail the following:

    1. 4 month's supply of Dapagliflozin
    2. A self-addressed envelope for return of the diary and pill bottles at the end of the dosing period
    3. A weighing scale (if required)
12. Dosing compliance will be checked during initial study treatment via sharing of pill accountability data or screenshot of paper pill diary
13. If clinically indicated, labs will be ordered and run more frequently to assess for toxicity.
14. Visits 3, 4, and 5 will be conducted in the same manner as described above.
15. All pill bottles and diaries (if paper version is used) will be returned via the provided envelope

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form.
* Stated willingness to comply with study procedures, including remote telehealth consultations with the study team, confirming availability, and agreeing to use mobile/web applications for study purposes.
* Age ≥18 years.
* Histopathologic diagnosis of renal AL amyloidosis confirmed by biopsy of any tissue and evidence of >1.0 g/day proteinuria without any other identifiable cause.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1 or 2.
* Plateau in any renal response (i.e., reduction in proteinuria) for at least 3 months prior to enrollment, as determined by the enrolling physician.
* Residence in the state of Michigan.

Exclusion Criteria:

* Either ongoing first line induction with anti-plasma cell therapy or ongoing post- induction maintenance for <6 months prior to enrollment.
* Diagnosis of symptomatic multiple myeloma, including presence of lytic bone disease, plasmacytomas, ≥60% plasma cells in the bone marrow, or hypercalcemia, either currently or in the past.
* Women of child-bearing potential (i.e., those who have not undergone chemical or surgical sterilization or are not postmenopausal) and who are unwilling to use a medically accepted and reliable form of contraception while participating in the study and for 2 weeks following the last dose of study medication, as determined by the investigator, or have a positive pregnancy test at the time of enrolment or are currently breastfeeding.
* Known allergic reactions to components of the dapagliflozin.
* Treatment requiring type 1 or type 2 diabetes mellitus.
* Baseline eGFR <25 mL/min/1.73m2.
* Acute or chronic liver disease with severe impairment of liver function (e.g., ascites, esophageal varices or coagulopathy)
* Current or previous use of any SGLT2i.
* Initiation or dose modification of angiotensin converting enzyme inhibitors (ACE inhibitors) and angiotensin receptor blockers (ARBs) <3 months prior to enrollment.
* Active malignancy requiring treatment (other than AL amyloidosis and non-melanoma skin cancers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving 30% reduction in daily proteinuria. | Up to Month 6
  A patient will be considered to have achieved the desired urine protein reduction if a 30% reduction in 24-hour albuminuria occurs at any point during the six-month period from the initiation of dapagliflozin therapy. The proportion of patients achieving this reduction will be calculated as the ratio of the total number of patients who experienced the reduction to the total number of evaluable patients.

SECONDARY OUTCOMES:
Completion rate of tele-visits | Up to Month 6
  The completion rate of tele-visits, including post-trial feedback, will be calculated as the ratio of completed tele-visits to scheduled tele-visits.

OTHER OUTCOMES:
Proportion of patients experiencing any of the following: (1) sustained decline in eGFR, (2) onset of ESRD, or (3) death from a renal disease-related or cardiovascular cause. | Up to Month 6
  A patient's status will be recorded as 'yes' if any of the following three events occur at any time during the 6 months of study therapy: a sustained ≥50% decline in estimated glomerular filtration rate (eGFR); the onset of dialysis-requiring end- stage renal disease (ESRD); or death from a renal disease-related or cardiovascular cause. Otherwise, the status will be marked as 'no'.
Incidence rate of developing dialysis dependent ESRD in patients with Pavia Renal AL Stage II or III involvement. | Up to Month 6
  The onset of ESRD in patients with Pavia Renal Stage II or III involvement will be recorded as binary (yes vs. no).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Zonder, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Karmanos Cancer Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No